CLINICAL TRIAL: NCT07236333
Title: The Role of CALLY and HAALP Scores in the Evaluation of Ulcerative Colitis Attack
Brief Title: The Role of CALLY and HAALP in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, okkes zortuk, Principal Investigator, Ataturk University
Other Study IDs: ZTKLAB30012025TBAEK121GASTROEN; TBAEK-121 (Other: Akdeniz University)
Record Dates: First submitted 2025-09-24; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; CALLY; HAALP
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CALLY — The CALLY index, integrating C-reactive protein (CRP), albumin, and lymphocyte count, has been identified as a promising prognostic biomarker.
Diagnostic Test: HALP — The HALP score is calculated as HALP Score = [hemoglobin (g/L) × albumin (g/L) × lymphocytes (/L)]/platelets (/L). It is a definitive biomarker.

SUMMARY:
The aim of this study is to demonstrate the type and amount of retention in the colon during ulcerative colitis activation, as well as the relationship between C-reactive protein (CRP), albumin and the calculated CALLY index. The investigators also aim to establish whether this ratio can be used to indicate activation.

ELIGIBILITY:
Inclusion Criteria:

* under 18

Exclusion Criteria:

* no UC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ulserative colitis patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Patients' HALP Score | through study completion, an average of 1 year
  Ulcerative colitis patients will be evaluated by evaluating the Change in HALP Score and its effect on prognosis.
Change in Patients' CALLY Index Score | through study completion, an average of 1 year
  Ulcerative colitis patients will be evaluated by evaluating the Change in CALLY Index Score and its effect on prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: 1. Further research on the clinical relevance of the ulcerative colitis colonoscopic index of severity for predicting 5-year relapse — http://doi.org/10.1007/S00384-021-04009-2
- See also: 2. Validation of a novel integral disease index for evaluating the grade of activity in Mexican patients with ulcerative colitis: A prospective cohort study — http://doi.org/10.1016/J.RGMXEN.2019.02.006